CLINICAL TRIAL: NCT03758027
Title: Communicate Alternatively, Release Endorphins, and Self-Soothe (CARESS) and Emotional Regulation for Cravings Management With Substance Use
Brief Title: CARESS: An Investigation of Effects of CARESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Principal Investigator, Maria Hadjiyane, Senior Director, Behavioral Health Adult Ambulatory Services, Inova Health Care Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #18-3023
Record Dates: First submitted 2018-09-27; First posted 2018-11-29 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Craving; Self Efficacy; Affective; Reaction; Substance Abuse
Keywords: emotional regulation; drug taking refusal skills; physiological responses
MeSH Terms: conditions — Substance-Related Disorders; Emotional Regulation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This will be a randomized control trial with an experimental and control group. There will be a total of 96 participants, 48 in each group. For research question, a 2 X 3 repeated measures MANOVA will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARESS (Experimental): The proposed intervention for this study has three stages: communicate alternatively (CA), release endorphins (RE), and self-soothe (SS) (CARESS)
  CARESS is a combined skill of three activities. Each section is timed and has specific activities:
  CA - will last eight (8) minutes, and will be expression of emotion with drawing with crayons.
  RE - will last six (6) minutes, and will be a butterfly hug with a blanket. SS - will last six (6) minutes, and will be a pre-recorded music selection.
  Interventions: Behavioral: CARESS
- ISOMETRIC (Active Comparator): This is a one time five-minute isometric circuit involving contracting muscles in different parts of the body. In order to be equivalent in time spent with the experimental intervention, this circuit will be performed three times with a five-minute break between each instance
  Interventions: Behavioral: Isometric Exercise

INTERVENTIONS:
Behavioral: CARESS — The goals of each component are as follows:
  * Communicate alternatively - a method to bring the brain back and remove the individual from his/her limbic system;
  * Release endorphins - a release for the internal stress created by the emotion; and
  * Self-soothe - a method of quelling and containing.
  Arms: CARESS
Behavioral: Isometric Exercise — 5-minute protocol for cravings management and affect regulation
  Arms: ISOMETRIC

SUMMARY:
The purpose of this research is to study the efficacy of an intervention that could interrupt the cycle of emotion dysregulation as it relates to cravings and negative emotions for those with problematic substance use behaviors. This will be a quantitative randomized control trial study with data collection at three points: pre-intervention, post-intervention, and same-day follow up. This study will be conducted at the Inova Behavioral Health Merrifield Center. Inova's addictions services program is the CATS program (formerly comprehensive addiction treatment services), which provides therapeutic interventions for those managing substance use disorders. The focus of measurement will be about the current state of the participant, and not a cumulative status. This one-session intervention. The goal is to have 96 participants in the study, 48 in each of the two groups.

DETAILED DESCRIPTION:
The conceptual framework for the study is built on a foundation of three models found in the literature. The first of these is Gross's model of emotional regulation (ER), a goal-oriented linear process allowing for interventions at different phases in the experience. The individual has choices to: (1) avoid a situation all together; (2) deflect or distract from the situation; (3) reframe the situation; (4) or manage the physiological reactions. Adding on to this model, Koole expanded the framework, and reclassified the processes as tasks toward a goal, while adding an array of functions for each task. This includes where he/she is focusing, what he/she is thinking, and how he/she is responding. This allows the individual more choices in managing the emotions, depending on what he/she is trying to achieve. Finally, applying a taxonomy developed by Webb et al. (2012) of interventions to this framework, the identification of types of interventions is clarified. The framework is then applied to the proposed intervention, CARESS.

The proposed study will investigate a specific intervention and its efficacy at managing the acute effects for cravings, drug and drinking refusal self-efficacy, physiological responses, and affect disturbance for those with problematic substance use behaviors. The intervention is a one-time treatment session using CARESS in comparison to a control group who do not receive CARESS for those with problematic substance use behaviors. The aim is to investigate the difference in variances between pre, post, and follow up measurements for cravings, drug and drinking refusal skill self-efficacy, affect disturbance, and physiological responses for a one-time treatment session using CARESS in comparison to a control group for those with problematic substance use behaviors.

This is the initial study with respect to CARESS overall

ELIGIBILITY:
Inclusion Criteria:

1. be 18 years or older
2. meet criteria for problematic drinking or drug use

Exclusion Criteria:

1. having been directly discharged from an inpatient psychiatric admission;
2. currently under the influence of alcohol or any illicit or non-prescribed drugs;
3. having received either of the treatment interventions as part of their current treatment;
4. having current suicidal or homicidal thoughts, plans, or attempts;
5. experiencing current psychosis; or
6. unable to read the self-report assessment forms in English without assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
Change in Cravings level | The single session is will last 2 hours, the intervention will last 20 minutes. The measures will be taken prior to the intervention, (pre-), immediately after the intervention, (post-), and 30 minutes after the conclusion (follow up).
  To identify the change in intensity and characteristics of cravings, using the Penn Alcohol Craving Scale (PACS). The Penn Alcohol Craving Scale (PACS) is a self-report tool addressing the frequency, intensity, and duration of craving, as well as the self-efficacy in the resistance to drink, and a comprehensive cravings measurement. Each question is on a Likert-scale with answers from zero (0) to six (6) and scores of questions one through four ranging from zero to 30, with no subscales. The lower the score the lower the craving, therefore a better outcome. The initial study of the PACS supported content, predictive and construct validity. There is an internal consistency of .92 Cronbach's alpha.

SECONDARY OUTCOMES:
Change in Affect disturbance | The single session is will last 2 hours, the intervention will last 20 minutes. The measures will be taken prior to the intervention, (pre-), immediately after the intervention, (post-), and 30 minutes after the conclusion (follow up).
  To identify the change in affect disturbance, the Positive Affect and Negative Affect Schedule (PANAS) instrument will be used. The PANAS is a 20-question instrument with 10 emotions listed for positive affect, and 10 emotions listed for negative affect. These are scored on a 5-point Likert scale, measuring the positive and negative affects an individual is experiencing at a specific moment in time. Although both scales are on the instrument, they do not measure the same continuum. The Positive affect subscale: questions 1, 3, 5, 9, 10, 12, 14, 16, 17, & 19, with scores ranging from 10 - 50; higher scores indicate more of a positive affect. The Cronbach's alpha for the positive affect subscale ranges from .86-.90. The Negative affect subscale: questions 2, 4, 6, 7, 8, 11, 13, 15, 18, & 20 with scores ranging from 10 - 50; lower scores indicate less of a negative affect. The Cronbach's alpha for the negative affect, a range of .84-.87.
Change in Physiological Responses | The single session is will last 2 hours, the intervention will last 20 minutes. The measures will be taken prior to the intervention, (pre-), immediately after the intervention, (post-), and 30 minutes after the conclusion (follow up).
  Identify the change in the galvanic skin response for the participant, utilizing GSR reader
Change in Drug taking refusal skills | The single session is will last 2 hours, the intervention will last 20 minutes. The measures will be taken prior to the intervention, (pre-), immediately after the intervention, (post-), and 30 minutes after the conclusion (follow up).
  Identify the change in perception of self-efficacy on drug refusal skills, utilizing Drug-Taking Confidence Questionnaire. The DTCQ-8 assesses a participant's confidence that he/she would not use drugs or drink in different scenarios of high-risk situations. The 8 questions each correspond to relapse predictors. Each item is scored on a scale of 0 to 100, in intervals of 20: 0, 0% not at all confident I would be able to resist; 20, 20% confidence to resist; 40, 40% confident; 60, 60% confident; 80, 80% confident; and 100, 100% very confident. There are two versions of the DTCQ-8, one for alcohol and one for drugs, the measurements are the same and the wording in the instructions is slightly different. It is recommended that the appropriate instrument be used for the drug of choice of the client. In order to score the full instrument, a global self-efficacy score is calculated by averaging the scored items; the higher the score, the greater the self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Hadjiyane, MA, MS, Principal Investigator — Sr. Director Behavioral Health Adult Ambulatory Services; Sylvia Marotta-Walters, PhD, Study Chair — Chair, Graduate School of Education and Human Development
Locations (1):
- Inova Behavioral Health, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No